CLINICAL TRIAL: NCT03960125
Title: Photodynamic Therapy and Microvesicles
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The PI decided to move in another direction with his research.
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 06714
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Photodynamic Therapy; Microvesicle Particle
MeSH Terms: interventions — Photochemotherapy; Imipramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 4% Imipramine Cream on Upper Forearm Site (Experimental): Base cream will be applied to the lower forearm site.
  Interventions: Device: Photodynamic Therapy; Drug: 4% Imipramine; Drug: Base Cream
- 4% Imipramine Cream on Lower Forearm Site (Experimental): Base cream will be applied to the upper forearm site.
  Interventions: Device: Photodynamic Therapy; Drug: 4% Imipramine; Drug: Base Cream

INTERVENTIONS:
Device: Photodynamic Therapy — Blue Light Therapy Exposure
Drug: 4% Imipramine — A tricyclic antidepressant (TCA) medication. Though it is usually taken orally, topical preparations (4%) has use in topical anesthetics and anti-pain medicaments.
Drug: Base Cream — Control to 4% Imipramine

SUMMARY:
This study is designed to test whether localized photodynamic therapy (PDT) treatment will result in increased skin levels of microvesicle particle (MVP) and if the use of imipramine will counteract PDT generated MVP release. The effects of PDT and ultraviolet B radiation (UVB) on platelet-activating factor (PAF) and MVP production have long been part of the PI's research experience. To test this, the investigator plans to enroll up to enroll up to 12 male subjects whom are aged 21 to age 45. These subjects will be treated with topical 5-aminolevulinic acid gel (Ameluz) to small areas of forearm followed by treatment with blue light. The areas will then be treated with either 4% imipramine cream or cream base as control. Four hours later, the redness of the areas will be measured using a mexameter and MVPs measured in skin biopsies taken from PDT-treated skin.

ELIGIBILITY:
Inclusion Criteria:

* Male adult subjects age 21 to age 45
* Skin type must be "fair", Fitzpatrick type I or II
* Able to understand/complete informed/consent
* Have access to stable transportation

Exclusion Criteria:

* Underlying diseases that could affect wound healing (e.g., diabetes mellitus)
* Taking medications that are known photosensitizers (e.g., doxycycline) or anti- inflammatories (e.g., NSAIDS [except for low-dose aspirin] or steroids)
* Have a history of abnormal scarring (e.g., keloids)
* Taking vitamin C or E supplements for past month
* Utilizing imipramine or any other tricyclic antidepressant (oral or cream)
* Utilizing topical anti-inflammatory or systemic agents (eg, prednisone)
* Tanning bed use within last 3 months
* PDT or UVB treatments in past 3 months

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Change in Microvesicle Particle Levels From Baseline with Photodynamic Therapy. | Day 0
  PI will assess change from baseline using three 5 mm punch biopsies.
Change in Microvesicle Particle Levels From Baseline with 4% Imipramine Cream Treatment. | Day 2
  PI will assess change from baseline using three 5 mm punch biopsies.

SECONDARY OUTCOMES:
Change in Erythema From Baseline Due to Photodynamic Therapy | Day 2
  PI will assess change from baseline by using a non-invasive mexameter.
Change in Skin Pain From Baseline Due to Photodynamic Therapy | Day 2
  PI will assess change with the Skin Pain Visual Analogue Scale. Participants indicate the overall severity of skin pain from the photodynamic therapy treatment at the present time by placing a single mark on the horizontal scale (0 = no skin pain to 10 = severe skin pain)
Change in Itch From Baseline Due to Photodynamic Therapy | Day 2
  PI will assess change with the Itch Numerical Scale. Participants will rate itching severity due to photodynamic therapy treatment by circling the number that best describes the worst level of itching in the past 24 hours. (0 = No itch to 10 = Worst itch imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Travers, MD, PhD, Principal Investigator — Wright State Physicians
Locations (1):
- Wright State Physicians, Fairborn, Ohio, United States

DOCUMENTS (1):
  • Informed Consent Form (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT03960125/ICF_000.pdf